CLINICAL TRIAL: NCT00200954
Title: Primary Prevention of Atopic Disease by Perinatal Administration of Probiotics.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Netherlands Asthma Foundation (Other)
Collaborators: UMC Utrecht (Other)
Responsible Party: M.O. Hoekstra, M.D., PhD., University Medical Centre Utrecht, Wilhelmina Childrens' Hospital, The Netherlands
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PANDA
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2008-08-18 (Estimated); Status verified 2007-05

CONDITIONS: Food Allergy; Atopic Dermatitis; Asthma; Rhinitis
Keywords: prospective; intervention; randomised; probiotics; atopy
MeSH Terms: conditions — Food Hypersensitivity; Dermatitis, Atopic; Asthma; Rhinitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- placebo (Placebo Comparator): placebo group
  Interventions: Dietary Supplement: Placebo
- 2 (Active Comparator): Probiotic bacteria group
  Interventions: Dietary Supplement: Probiotic bacteria

INTERVENTIONS:
Dietary Supplement: Probiotic bacteria — 3 x 10e9 CFU of a mixture of probiotic bacteria, once daily to the pregnant mothers last 6 weeks of pregnancy.To their offspring during the first year of life.
  Arms: 2
Dietary Supplement: Placebo — The placebo consists of the carrier of the probiotic bacteria mixture, i.e. rice starch and maltodextran
  Arms: placebo

SUMMARY:
Administration of probiotics to pregnant women from an atopic family and subsequently to their high-risk newborns results in prevention of the incidence or in a decrease of the severity of atopic disease during infancy.

DETAILED DESCRIPTION:
Background. Atopic diseases are increasing in countries with a Western lifestyle. The hygiene hypothesis states that the increase in atopic disease could be due to reduced exposure to microbial antigens in early in life. In search of new preventive therapies for atopic disease, exposure of pregnant women with previous or recent atopic disease, and their offspring to probiotics has been suggested. Probiotics are mono or mixed cultures of microbes which, when applied to animal or man, can beneficially affect the host, among others by inducing an immune response. Probiotics are generally accepted to be safe in children. Probiotics have shown to be effective in primary prevention of atopic disease in high-risk neonates in one study so far. However, it is still unclear by what mechanism probiotics work and which is the most immunopotent (combinations of) probiotic(s). It is likely that antigen-presenting cells (APC's) are involved, since these cells are important in the first line of defence in the gastrointestinal tract. It can be imagined that the immune response is the result of the interplay between probiotics and APC's. In particular, the match between pathogen-associated molecular patterns (PAMP's) on probiotics and their counterparts on APC's, the pathogen-recognition-receptors (PRR's) (like for instance Toll-like receptors) is decisive in this aspect.

Hypothesis. Administration of probiotics to pregnant women and their offspring may reduce the development of sensitization as well as the onset of atopic disease in their offspring.

Aim. To study the effect of probiotics on sensitisation and the prevalence of atopic disease, the severity of atopic disease, the intestinal flora and immune parameters in high-risk newborns.

Methods. To study this hypothesis, a randomised, double-blind placebo-controlled trial will be carried out by administration of probiotics to pregnant women with previous or recent atopic disease as well as to their offspring. Primary outcome parameters are firstly the prevalence and severity of sensitization and atopic disease in the offspring during a follow-up of two years. Secondary outcome parameters are the change in stool composition during treatment with probiotics and in-vitro production of cytokines by PBMCs collected at 3 months, 1 year and 2 years of age.

Expected results. Perinatal administration of probiotics to pregnant women and their offspring may hamper the development of sensitization and atopic disease in their offspring. This may be due to modulation of the intestinal microbiota composition, and modulation of the developing immune system

ELIGIBILITY:
Inclusion Criteria:

* Pregnant mothers were included if either they themselves or their husband plus one sibling suffered from present or past atopic disease

Exclusion Criteria:

* Maternal use of immunomodulatory drugs during pregnancy, the use of probiotics prior to the start of the study.
* Children were excluded from the study if their mother received antibiotic treatment during the last two weeks of pregnancy
* When the child was born preterm, i.e. before 37 weeks of gestation
* If the children received antibiotic treatment in the first two weeks of life
* If ingestion of the study product was difficult due to vomiting or feeding problems in general for longer than 3 weeks from birth
* If the children had other major medical problems

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 157 (Actual)
Dates: Start 2004-01; Primary Completion 2007-12 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of atopic disease at the age of 2 years. Incidence and prevalence of eczema | Follow-up at 3 months, 12 months, and 24 months

SECONDARY OUTCOMES:
Serum IgE, stool composition, cytokines produced by PBMNC's | Follow-up at 3 months, 12 months and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Maarten O Hoekstra, MD PhD, Principal Investigator — Wilhelmina Children's Hospital Utrecht (UMCU)
Locations (1):
- Wilhelmina Children's Hospital (UMCU), Utrecht, Utrecht, Netherlands

REFERENCES:
- See also: Related Info — http://www.kinderallergologie.nl